CLINICAL TRIAL: NCT06559917
Title: Effectiveness on Family Cohesion and Happiness of Using Social Media to Enhance Happiness Accounts for Late-Stage Cancer Patients and Their Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YANG WEN-CHI (Other)
Responsible Party: Sponsor-Investigator, YANG WEN-CHI, Graduate Student in Nursing, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: A202405117
Record Dates: First submitted 2024-08-06; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Upon admission to the cancer-related ward, after explaining the purpose and process of the study, patients who agree to participate in the study will complete the first questionnaire before the intervention with the social media "Happiness Ledger". The family members will have one week to organize photos, after which the patients will share the meaning of the photos. The process will be recorded by the researcher and will last approximately 40 to 60 minutes. Afterward, the researcher will create a video of about three minutes using the photos and ask the participating family members to assist in uploading the photos to the family LINE group as feedback to the research subjects. The patients will then complete the second questionnaire.
  Interventions: Other: life review
- Control Group (No Intervention): After explaining the purpose and process of the study to the patients and their family members on the day of admission, and obtaining their consent to participate in the study, they will complete the first questionnaire. One week later, they will complete the second questionnaire. After the entire study is completed, the control group will receive the same social media "Happiness Ledger" intervention as the experimental group. Data collection will be conducted for both groups before and after the intervention.

INTERVENTIONS:
Other: life review — After consenting, they will complete the first questionnaire before receiving the "Happiness Ledger" intervention via social media. Family members will have one week to organize photos, after which patients will share the meaning of the photos. This process will be recorded by the researcher and will last approximately 40 to 60 minutes. The researcher will then create a three-minute video using the photos, and the participating family members will assist in uploading the photos to the family LINE group as feedback to the subjects. The second questionnaire will then be completed.
  Arms: Experimental Group

SUMMARY:
The study period is from September 1, 2024, to December 31, 2025. The subjects are cancer patients from the medical center of this hospital. A block randomization will be used to assign 100 patients to the experimental group and 100 patients to the control group, totaling 200 patients. During the study process, questionnaires and medical records of the subjects will be collected. The experimental group will receive the social media "Happiness Ledger" intervention, while the control group will receive routine treatment. Questionnaires will be collected from both groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria for Advanced Cancer Patients:

1. Patients diagnosed with stage III or IV cancer by a specialist physician.
2. Patients who agree to participate in the study after being informed about the research.
3. Patients who are conscious and able to communicate in Mandarin or Taiwanese.
4. Patients aged 20 years or older.
5. Patients with no history of mental illness.

Inclusion Criteria for Family Members:

1. The primary caregiver of a patient diagnosed with stage III or IV cancer by a specialist physician.
2. The primary caregiver who has a blood, marital, or cohabitation relationship with the patient.
3. Family members who agree to participate in the study after being informed about the research.
4. Family members who are conscious and able to communicate in Mandarin or Taiwanese.
5. Family members aged 20 years or older.
6. Family members with no history of mental illness.

Exclusion Criteria:

-

Exclusion Criteria for Advanced Cancer Patients:

1. Patients in the experimental group and control group who reside in the same ward.
2. Patients who share a ward with subjects already included in the study.
3. Patients involved in ongoing medical disputes.
4. Patients who cannot understand the study explanation due to language or cognitive impairments.
5. Patients with a life expectancy shorter than the planned study duration.

Exclusion Criteria for Family Members:

1. Family members who do not have direct living or caregiving contact with the patient.
2. Family members who cannot visit the patient regularly or participate in the study.
3. Family members who cannot understand the study explanation due to language or cognitive impairments.
4. Family members with significant visual or hearing impairments who do not use assistive devices and cannot resolve communication issues.
5. Family members who cannot make independent decisions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Family Cohesion | Baseline (pre-intervention) and 1 week after intervention
  This study uses the Family Adaptability and Cohesion Evaluation Scale (FACES II) developed by Olson et al. (1979), which consists of 30 items to measure the family cohesion of patients and their families .

SECONDARY OUTCOMES:
Happiness | Baseline and 1 week
  This study uses the Subjective Happiness Scale (SHS) created by Lyubomirsky & Lepper (1999), which consists of 4 items to measure the happiness of patients and their families."

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang WC, Li CY, Ho CL, Chang PY, Wu LF, Pan HH. Effectiveness of a Social Media-Based Life Review Intervention on Happiness in Advanced Cancer Patients and Their Family Caregivers: A Mixed-Methods Study. Psychooncology. 2026 Jan;35(1):e70374. doi: 10.1002/pon.70374. PMID 41478730